CLINICAL TRIAL: NCT00936156
Title: Treatment of High-Risk Cerebral Primitive Neuroectodermal Tumors in Children Aged Over 5 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PNET HR+ 5; CSET 1329
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Metastatic, Cerebral Primitive Neuroectodermal Tumors
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Drug Therapy; Carboplatin; Etoposide; Thiotepa

ARMS (1):
- Chemotherapy (Experimental): Conventional chemotherapy: carboplatin injection (160 mg/m²/day by infusion over one hour in 5 % glucose saline) administered from D1 to D5 and from D22 to D26. Etoposide injection (100 mg/m²/day by infusion over one hour in 5 % glucose saline) administered from D1 to D5 and from D22 to D26. Double intensification by high-dose chemotherapy followed by autologous PBSC rescue: thiotepa injection (200 mg/m²/day as an infusion over one hour in 200 ml/m² of 5 % GS) administered from D42 to D44 and from D63 to D65. Autologous PBSC rescue on D47 and D68. Surgical resection of any tumor residue. Irradiation of the primary tumor site and cerebrospinal axis: 54 Gy to primary tumor, 36 Gy to cerebrospinal axis. Maintenance treatment: Temozolomide 150 mg/m²/day orally for 5 days every 28 days, from 1 month after the end of irradiation. 6 cycles planned. Duration of treatment: 13 months
  Interventions: Drug: Chemotherapy (carboplatin, etoposide, thiotepa)

INTERVENTIONS:
Drug: Chemotherapy (carboplatin, etoposide, thiotepa) — Conventional chemotherapy: carboplatin injection (160 mg/m²/day by infusion over one hour in 5 % glucose saline) administered from D1 to D5 and from D22 to D26. Etoposide injection (100 mg/m²/day by infusion over one hour in 5 % glucose saline) administered from D1 to D5 and from D22 to D26. Double intensification by high-dose chemotherapy followed by autologous PBSC rescue: thiotepa injection (200 mg/m²/day as an infusion over one hour in 200 ml/m² of 5 % GS) administered from D42 to D44 and from D63 to D65. Autologous PBSC rescue on D47 and D68. Surgical resection of any tumor residue. Irradiation of the primary tumor site and cerebrospinal axis: 54 Gy to primary tumor, 36 Gy to cerebrospinal axis. Maintenance treatment: Temozolomide 150 mg/m²/day orally for 5 days every 28 days, from 1 month after the end of irradiation. 6 cycles planned. Duration of treatment: 13 months

SUMMARY:
Primary objective : To increase the 3 year progression-free survival from 40% to 60%. Patients included : metastatic, cerebral primitive neuroectodermal tumors in children aged over 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Type of tumor:

   * Metastatic medulloblastoma whatever the quality of the initial resection (radiologically visible metastases by MRI and/or CSF invaded by at least one mass of tumoral cells).
   * Incompletely resected local medulloblastoma with a residue > 1.5 cm2.
   * Anaplastic, large cell medulloblastoma whatever the risk criteria (localized or metastatic, complete or incomplete resection).
   * Medulloblastoma with amplification of c-myc or N-myc whatever the risk criteria (local or metastatic, complete or incomplete resection).
   * Local and/or metastatic sustentorial PNET.
2. Age at diagnosis of the medulloblastoma of more than 5 years and less than 20 years.
3. Age at diagnosis of S-PNET of more than 10 years and less than 20 years.
4. Nutritional and general status compatible with treatment, Lansky score > 60.
5. Estimated life expectancy > 1 months.
6. Radiographs must be available for the second reading in dicom format on a CD-ROM.
7. Hematological function at diagnosis: PMN > 1.0 x 109/l and platelets > 100 x 109/l.
8. Hepatic function at diagnosis: serum bilirubin < 1.5 times normal value; ASAT and ALAT < 2.5 times normal values; prothrombin time > 50%; fibrinogen > 1.5 g/l.
9. Renal function at diagnosis: serum creatinine according to age in a correctly hydrated child: 1 to 15 years < 65 micromol/l; 15 to 18 years < 110 micromol/l.
10. No organ toxicity (Grade > 2 according to NCI-CTC coding, version 2.0)
11. No other concomitant anti-cancer treatment.
12. No prior anti-cancer therapy.
13. No prior irradiation.
14. Written informed consent signed by both parents or legal guardians

Exclusion Criteria:

1. Failure to comply with one of the inclusion criteria.
2. Severe or life-threatening infection.
3. Uncontrolled active or symptomatic intracranial hypertension.
4. Refusal of parents or legal guardian.
5. Patients incapable of undergoing medical follow-up for geographical, social or mental reasons

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2009-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Gustave Roussy, Villejuif, France

REFERENCES:
- [Derived] Larrouquere L, Dufour C, Faure-Conter C, Alapetite C, Meyronet D, Bolle S, Bonneville-Levard A, Sunyach MP, Laurence V, Frappaz D. Intensive pediatric chemotherapy regimen (PNET HR+5) in adult high-risk medulloblastoma and pineoblastoma patients. Neurooncol Adv. 2024 Aug 10;6(1):vdae141. doi: 10.1093/noajnl/vdae141. eCollection 2024 Jan-Dec. PMID 39620201
- See also: Related Info — http://www.igr.fr/